CLINICAL TRIAL: NCT03684044
Title: A Phase III, Randomized, Double-Blind Placebo-Controlled, Multicenter Study To Evaluate the Efficacy and Safety of Baloxavir Marboxil in Combination With Standard-of-Care Neuraminidase Inhibitor in Hospitalized Participants With Severe Influenza
Brief Title: Study to Assess Efficacy and Safety of Baloxavir Marboxil In Combination With Standard-of-Care Neuraminidase Inhibitor In Hospitalized Participants With Severe Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP40617; 2018-001416-30 (EudraCT Number)
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Results first posted 2020-11-30 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baloxavir Marboxil (Experimental): Participants will receive at least two doses of baloxavir marboxil on Days 1 and 4. A third dose of Baloxavir will be given on Day 7 for participants who have not improved according to protocol defined criteria on Day 5.
  Study treatment will be given in combination with SOC NAI (i.e., oseltamivir, zanamivir, or peramivir) in accordance with local clinical practice.
  Interventions: Drug: Baloxavir Marboxil
- Placebo (Placebo Comparator): Participants will receive at least two doses of placebo on Day 1 and 4. A third dose of placebo will be given on Day 7 for participants who have not improved according to protocol defined criteria on Day 5.
  Study treatment will be given in combination with SOC NAI (i.e., oseltamivir, zanamivir, or peramivir) in accordance with local clinical practice.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Baloxavir Marboxil — Baloxavir marboxil will be administered as a weight-based dose on Days 1 and 4. A third dose will be given on Day 7 for participants who have not improved according to protocol defined criteria on Day 5.
  Arms: Baloxavir Marboxil
Other: Placebo — Participants will receive matching placebo on Days 1, 4 and 7.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of baloxavir marboxil in combination with a standard-of-care (SOC) neuraminidase inhibitor (NAI) (i.e., oseltamivir, zanamivir, or peramivir) compared with a matching placebo in combination with a SOC NAI in hospitalized patients with influenza.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants: Signed informed consent by any participant capable of giving consent, or, where the participant is not capable of giving consent, by his or her legal/authorized representative
* Adolescent participants not able to legally consent: written informed consent for study participation is obtained from participant's parents or legal guardian, with assent as appropriate by the participant, depending on the participant's level of understanding and capability to provide assent
* Participants who require hospitalization for severe influenza or acquire influenza during hospitalization, the severity of which requires an extension of hospitalization
* Diagnosis of influenza A and/or B by a positive Rapid Influenza Diagnostic Test (RIDT) or reverse transcriptase-polymerase chain reaction (RT-PCR)
* The time interval between the onset of symptoms and randomization is within 96 hours
* A score of ≥4 based on the National Early Warning Score 2 (NEWS2)
* Participants will require objective criteria of seriousness defined by at least one of the following criteria:
* Requires ventilation or supplemental oxygen to support respiration
* Has a complication related to influenza that requires hospitalization (e.g., pneumonia, central nervous system involvement, myositis, rhabdomyolysis, acute exacerbation of chronic kidney disease, asthma or chronic obstructive pulmonary disease (COPD), severe dehydration, myocarditis, pericarditis, exacerbation of ischemic heart disease)
* For women of childbearing potential: Agreement to remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 28 days after the last dose of study treatment. Hormonal contraceptive methods must be supplemented by a barrier method.

Exclusion Criteria:

* Participants who have received more than 48 hours of antiviral treatment for the current influenza infection prior to screening
* Participants who have received baloxavir marboxil for the current influenza infection
* Known contraindication to neuraminidase inhibitors
* Participants hospitalized for exclusively social reasons (e.g., lack of caregivers at home)
* Participants expected to die or be discharged within 48 hours, according to the investigator's judgement
* Participants weighing < 40 kg
* Participants with known severe renal impairment (estimated glomerular filtration rate < 30 mL/min/1.73 m2) or receiving continuous renal replacement therapy, hemodialysis, peritoneal dialysis
* Participants with any of the following laboratory abnormalities detected within 24 hours prior to or during screening (according to local laboratory reference ranges:
* Alanine Transaminase (ALT) or Aspartate Transaminase (AST) level > 5 times the upper limit of normal (ULN) OR
* ALT or AST > 3 times the ULN and total bilirubin level > 2 times the ULN
* Pregnant or breastfeeding, or positive pregnancy test in a predose examination, or intending to become pregnant during the study or within 28 days after the last dose of study treatment
* Exposure to an investigational drug within 5 half-lives or 30 days (whichever is longer) of randomization
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study
* Known hypersensitivity to baloxavir marboxil or the drug product excipients

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (170):
- United States (14):
  - Torrance Memorial Medical Center, Torrance, California
  - Denver Health Medical Center, Denver, Colorado
  - Atlanta Institute For Medical Research, Inc; DeKalb Medical Pharmacy, Decatur, Georgia
  - University of Chicago; Oncology Dept, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Barnum Medical Research, Inc., Natchitoches, Louisiana
  - Detroit Receiving Hospital, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - Creighton University Medical Center, Omaha, Nebraska
  - New York-Presbyterian Brooklyn Methodist Hospital; Department of Emergency Medicine, Brooklyn, New York
  - Temple University Hospital ; Lung Center, Philadelphia, Pennsylvania
  - Salem Veterans Affairs Medical Center - NAVREF; Pharmacy, Salem, Virginia
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Instituto Medico Platense, La Plata, Argentina
- Australia (2):
  - Royal Brisbane & Womens Hospital; Pharmacy Department, Herston, Queensland
  - Royal Children's Hospital Melbourne - PIN, Parkville, Victoria
- Belgium (3):
  - Hopital Erasme; Chest Medicine, Cardiac & Thoracic Surgery, Brussels
  - Cliniques Universitaires Saint-Luc; Hematology, Brussels
  - UZ Leuven, Leuven
- Brazil (3):
  - Santa Casa de Misericordia; de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Centro de Estudos Clinicos do Interior Paulista, Jaú, São Paulo
- Bulgaria (14):
  - Multiprofile Hospital For Active Treatment Sveta Ekaterina Dimitrovgrad EOOD; Internal Diseases, Dimitrovgrad
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases - Haskovo EOOD, Haskovo
  - MHAT Stamen Iliev AD; Pharmacy, Montana
  - University Mulitiprofile Hospital for Active Treatment Sveti Georgi EAD; Pharmacy, Plovdiv
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases Dr. D. Gramatikov - Ruse, Rousse
  - Multiprofile Hospital for Active Treatment - Samokov EOOD, Samokov
  - Multiprofile Hospital For Active Treatment Sliven То Military Hospital Sofia; Pharmacy, Sliven
  - Multiprofile Hospital For Active Treatment - Dr. Bratan Shukerov AD; Pharmacy, Smolyan
  - First Multiprofile Hospital for Active Treatment - Sofia EAD, Sofia
  - Fifth Multiprofile Hospital for Active Treatment - Sofia EAD; Pharmacy, Sofia
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia; Pharmacy, Sofia
  - National Multiprofile Transport Hospital Tzar Boris Ill; Clinic of Internal Diseases, Sofia
  - Multiprofile District Hospital for Active Treatment Dr. Stefan Cherkezov AD; Pharmacy, Veliko Tarnovo
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases-Vratsa; Pharmacy, Vratsa
- Canada (8):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Carlson Urology, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Toronto East General Hospital; Main Pharmacy G Wing Basement, East York, Ontario
  - London Health Sciences Center; Pharmacy Dept., London, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie, Québec
- China (10):
  - Beijing Ditan Hospital Capital Medical University, Beijing
  - Beijing Youan Hospital, Capital Medical University; Center for Infectious Diseases, Beijing
  - China-Japan Friendship Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - Ruijin Hospital (GuangCi Hospital), Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
- Czechia (2):
  - Fakultni nemocnice Brno; Interni hematologicka a onkologicka klinika, Brno
  - Nemocnice Kyjov, prispevkova organizace, Kyjov
- East Tallinn Central Hospital, Tallinn, Estonia
- Finland (3):
  - Kuopion Yliopistollinen Sairaala; Silmätaudit, Kuopio
  - Oulun Yliopistollinen Sairaala; Teho-osasto, Oulu
  - Turku University Hospital, Turku
- France (10):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - CHRU Dijon Complexe Du Bocage, Dijon
  - Centre Hospitalier Departemental de Vendee, La Roche-sur-Yon
  - Hôpital Universitaire Dupuytren, Limoges
  - CHRU Nantes, Nantes
  - CHU de Nîmes - Hôpital Carémeau, Nîmes
  - Hopital de La Source, Orléans
  - Groupe Hospitalier Pitie Salpetriere; Service De Pneumologie, Paris
  - Nouvel Hopital Civil - CHU Strasbourg, Strasbourg
  - CHRU Bretonneau, Tours
- Germany (9):
  - Uniklinik Koln; Klinik I fur Innere Medizin, Cologne
  - Krankenhaus Donaustauf der LVA Niederbayern Oberpfalz, Donaustauf
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - St. Josefskrankenhaus - Freiburg; Klinik fur Pneumologieund Beatmungsmedizin, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Schleswig-Holstein; Klinik fuer Innere Medizin I, Lübeck
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Klinikum der Universität Regensburg, Regensburg
  - Universitatsklinikum Tubingen, Tübingen
- Hong Kong (3):
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin, New Territories
- Israel (8):
  - Soroka University Medical Centre, Beersheba
  - Edith Wolfson Medical Center, Holon
  - Galilee Medical Center, Nahariya
  - Chaim Sheba Medical Center; Allergy and Clinical Immunology Unit, Ramat Gan
  - Rambam Health Corporation; Oncology Institute, Rambam
  - ZIV Medical Center; Department Of Internal Medicine A, Safed
  - Tel Aviv Sourasky Medical Center; Pharmacy, Tel Aviv
  - Baruch Padeh Poria Medical Center; Pharmacy, Tiberias
- Japan (19):
  - Fujita General Hospital, Dategun Kunimimachi
  - Shin Komonji Hospital, Fukuoka
  - Fukuoka Shin Mizumaki Hospital, Fukuoka
  - Fukuoka Wajiro Hospital, Fukuoka
  - Rinku General Medical Center, Izumisano
  - National Hospital Organization Minami Kyoto Hospital, Jōyō
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Naha City Hospital, Naha
  - National Hospital Organization Ibarakihigashi National Hospital; Center for Clinical Research, Naka-gun
  - Japan Community Health care Organization Nihonmatsu hospital, Nihonmatsu
  - Social Corporation Keigakukai Minamiosaka Hosupital, Osaka
  - National Hospital Organaization Shibukawa Medical Center, Shibukawa
  - Tokyo Shinagawa Hospital Medical Corporation Association Tokyokyojuno-kai, Shinagawa City
  - Saka General Hospital, Shiogama
  - Local incorporated administrative agency Shizuoka City Shizuoka Hospital, Shizuoka
  - Iwase General Hospital, Sukagawa
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
  - Nagata Hospital; Department of pulmonary medicine, Yanagawa-shi
- Mexico (4):
  - Instituto Nacional de Ciencias Médicas y Nutricion Dr. Salvador Zubiran; Hamatologia y Oncologia, México, Mexico CITY (federal District)
  - Hospital Civil Fray Antonio Alcalde; Instituto de Patologia Infecciosa, Guadalajara
  - Hospital Universitario Dr. Jose Eleuterio González; Enfermedades Pulmonares Crónicas, Monterrey
  - Hospital General de Tijuana, Tijuana
- Netherlands (5):
  - Leids Universitair Medisch Centrum; C5-P Stafcentrum Hartziekten, Leiden
  - Canisius Wilhelmina Ziekenhuis; Department Hematology, Nijmegen
  - Ikazia Ziekenhuis, Rotterdam
  - Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Wellington Hospital, Wellington, New Zealand
- Peru (2):
  - Hospital Alberto Sabogal Sologuren, Callao
  - Hospital Nacional Adolfo Guevara Velasco - ESSALUD; Servicio de Cardiología, Cusco
- Romania (7):
  - Prof. Dr. Matei Bals Institute of Infectious Diseases, Bucharest
  - Dr. Victor Babes Clinical Hospital For Tropical and Infectious Diseases, Bucharest
  - Spitalul Clinic de Boli Infectioase, Cluj-Napoca
  - Sf.Cuv. Parascheva Infectious Diseases Clinical Hospital, Galati
  - Spitalul Clinic de Boli Infectioase "Sfanta Parascheva" Iasi, Iași
  - Sibiu Emergency Clinical County Hospital, Sibiu
  - Sf. Ioan cel Nou Emergency County Hospital, Suceava
- Serbia (7):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - Institute of Lung Diseases Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis; Clinic for Pulmonary Diseases and Tuberculosis Knez Selo, Niš
  - Clinical Centre of Vojvodina, Nova Sad
  - General Hospital Dr Radivoj Simonovic Sombor, Sombor
- Tan Tock Seng Hospital, Singapore, Singapore
- South Korea (7):
  - The Catholic University of Korea Incheon St. Mary's Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - ChungAng University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (12):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Joan de Deu - PIN; Unitat de Recerca - Farmacia, Esplugues de Llobregat, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Hospital General Universitario Reina Sofia; Servicio de Nefrologia, Murcia
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital de La Ribera, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skånes Universitetssjukhus Malmö; Infektionskliniken, Malmo
- Turkey (Türkiye) (4):
  - Hacettepe University Medical Faculty, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Selcuk University Medical Faculty; Internal Medicine, Konya
  - Karadeniz Technical University Faculty of Medicine, Trabzon
- Ukraine (8):
  - Regional Municipal Institution Chernivtsi Regional Clinical Hospital, Chernivtsi, Chernihiv Governorate
  - Kyiv Oleksandrivska Clinical Hospital; Infectious Box Department #2, Kyiv, Katerynoslav Governorate
  - Regional Municipal Institution Sumy Regional Infectious Clinical Hospital n.a. Z.Y. Krasovytskyi, Sumy, Katerynoslav Governorate
  - Ternopil City Municipal Emergency Hospital; Infectious Department, Ternopil, KIEV Governorate
  - Communal Non-Commercial Enterprise "Vinnytsia City Clinical Hospital №1"; Infectious Department, Vinnytsia, KIEV Governorate
  - MI Vinnytsia Regional Clinical Children's Infectious Hospital; Infectiuos Box department, Vinnytsia, KIEV Governorate
  - MI Dnipropetrovsk City Clinical Hospital #21 n.a. Prof. Popkova of DRC; The First Department, Dnipro, Podolia Governorate
  - Municipal Institution City Clinical Infectious Diseases Hospital, Odesa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Stannard HL, Mifsud EJ, Wildum S, Brown SK, Koszalka P, Shishido T, Kojima S, Omoto S, Baba K, Kuhlbusch K, Hurt AC, Barr IG. Assessing the fitness of a dual-antiviral drug resistant human influenza virus in the ferret model. Commun Biol. 2022 Sep 28;5(1):1026. doi: 10.1038/s42003-022-04005-4. PMID 36171475
- [Derived] Kumar D, Ison MG, Mira JP, Welte T, Hwan Ha J, Hui DS, Zhong N, Saito T, Katugampola L, Collinson N, Williams S, Wildum S, Ackrill A, Clinch B, Lee N. Combining baloxavir marboxil with standard-of-care neuraminidase inhibitor in patients hospitalised with severe influenza (FLAGSTONE): a randomised, parallel-group, double-blind, placebo-controlled, superiority trial. Lancet Infect Dis. 2022 May;22(5):718-730. doi: 10.1016/S1473-3099(21)00469-2. Epub 2022 Jan 24. PMID 35085510
- [Derived] Young B, Tan TT, Leo YS. The place for remdesivir in COVID-19 treatment. Lancet Infect Dis. 2021 Jan;21(1):20-21. doi: 10.1016/S1473-3099(20)30911-7. Epub 2020 Nov 26. No abstract available. PMID 33248473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 363 patients received at least one dose of study treatment and were included in the analyses of safety and efficacy.
Groups:
- Baloxavir Marboxil: Participants will receive at least two doses of baloxavir marboxil on Days 1 and 4. A third dose of Baloxavir will be given on Day 7 for participants who have not improved according to protocol defined criteria on Day 5. Study treatment will be given in combination with standard of care (SOC) NAI (i.e., oseltamivir, zanamivir, or peramivir) in accordance with local clinical practice.
Period: Overall Study
Arm/Group | Baloxavir Marboxil | Placebo
Started | 239 | 124
Completed | 217 | 104
Not Completed | 22 | 20
Not completed — Adverse Event | 3 | 0
Not completed — Death | 4 | 7
Not completed — Lost to Follow-up | 3 | 2
Not completed — Patient Not Available | 0 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baloxavir Marboxil | Placebo | Total
Number analyzed (Participants) | 239 | 124 | 363
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (19.8) | 61.6 (20.3) | 59.2 (20.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 56 | 173
  Male | 122 | 68 | 190
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 16 | 46
  Not Hispanic or Latino | 203 | 106 | 309
  Not Stated | 4 | 1 | 5
  Unknown | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 39 | 22 | 61
  Black or African American | 7 | 2 | 9
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White | 181 | 95 | 276
  Unknown | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinical Improvement
Description: Time to Clinical Improvement (TTCI) is defined as Time to Hospital Discharge OR Time to NEWS2 (National Early Warning Score 2) of ≤ 2 maintained for 24 hours.
Time Frame: Up to Day 35
Population: Participants were reverse transcriptase-polymerase chain reaction (RT-PCR) positive for influenza at any time point
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
hours | 97.5 [75.9 to 117.2] | 100.2 [75.9 to 144.4]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p = 0.4666, Gehan Wilcoxon; The Gehan Wilcoxon test was used to analyze the TTCI data because the proportional hazards assumption was violated; Median Difference (Net) = -2.7, 95% CI 2-sided [-53.4 to 25.9]

2. Secondary Outcome: Response Rates of the 6-Point Ordinal Scale at Day 7
Description: The ordinal scale categories are:
  Category 1) Discharged (or "ready for discharge") Category 2) Non-ICU hospital ward (or "ready for hospital ward") not requiring supplemental oxygen/non-invasive ventilation Category 3) Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen/non-invasive ventilation Category 4) ICU without mechanical (invasive) ventilation (or "ready for ICU admission") Category 5) Mechanical (invasive) ventilation Category 6) Death
Time Frame: Day 7
Population: All participants who were RT-PCR positive for influenza and were not discontinued or lost to follow up prior to day 7.
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 199 | 108
percentage of participants
  Category 1 | 49.2 | 45.4
  Category 2 | 22.6 | 24.1
  Category 3 | 20.1 | 22.2
  Category 4 | 4.0 | 1.9
  Category 5 | 3.5 | 4.6
  Category 6 | 0.5 | 1.9
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p = 0.6326, Cochran-Mantel-Haenszel; Statistic was stratified by region, NEWS2 at baseline (≤7, >7), and time from symptom onset to study treatment (≤48 hours, >48 hours)

3. Secondary Outcome: Time to Clinical Response
Description: Time to Clinical Response is based on temperature ranges, oxygen saturation, respiratory status, heart rate, and hospitalization status.
Time Frame: Up to Day 35
Population: Participants were RT-PCR positive for influenza at any time point
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
hours | 138.3 [120.0 to 161.1] | 145.1 [128.0 to 187.2]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p = 0.3272, Gehan Wilcoxon; The Gehan Wilcoxon test was used to analyze the TTCI data because the proportional hazards assumption was violated; Mean Difference (Net) = -6.8, 95% CI 2-sided [-50.9 to 17.7]

4. Secondary Outcome: Percentage of Participants on Mechanical Ventilation
Time Frame: Up to Day 35
Population: Participants were RT-PCR positive for influenza at any time point
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
percentage of participants | 5.3 | 6.1

5. Secondary Outcome: Duration of Mechanical Ventilation
Time Frame: Up to Day 35
Population: Participants were RT-PCR positive for influenza at any time point
Measure: Median (Full Range); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
hours | 150.25 [18.0 to 465.0] | 91.00 [24.0 to 407.0]

6. Secondary Outcome: Percentage of Participants Requiring ICU Stay
Time Frame: Up to Day 35
Population: Participants were RT-PCR positive for influenza at any time point
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
percentage of participants | 4.3 | 3.5

7. Secondary Outcome: Duration of ICU Stay
Time Frame: Up to Day 35
Population: Participants were RT-PCR positive for influenza at any time point
Measure: Median (Full Range); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
hours | 138.55 [23.7 to 362.0] | 71.78 [18.7 to 139.4]

8. Secondary Outcome: Time to Clinical Failure
Description: Time to clinical failure, defined as the time to death, mechanical ventilation, or ICU admission, corresponding to ordinal scale categories 6, 5, and 4, respectively, from baseline
Time Frame: Up to Day 35
Population: Participants were RT-PCR positive for influenza at any time point
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
hours | NA [NA to NA] — Very few patients experienced a clinical failure event and the median time to clinical failure could not be estimated . | NA [NA to NA] — Very few patients experienced a clinical failure event and the median time to clinical failure could not be estimated .

9. Secondary Outcome: Time to Hospital Discharge
Time Frame: Up to Day 35
Population: Participants were RT-PCR positive for influenza at any time point
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
hours | 166.7 [144.7 to 190.7] | 167.3 [146.4 to 211.1]

10. Secondary Outcome: Percentage of Participants With Post-Treatment Influenza-Related Complications
Description: Influenza-related complications included pneumonia, myositis or rhabdomyolysis, encephalitis or encephalopathy, myocarditis and/or pericarditis, otitis media, sinusitis, exacerbation of COPD/asthma, sepsis, acute lung injury or acute respiratory distress syndrome.
Time Frame: Up to Day 35
Population: Participants were RT-PCR positive for influenza at any time point
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
percentage of participants | 10.6 | 14.0

11. Secondary Outcome: Mortality Rate at Day 7
Time Frame: Up to Day 7
Population: Participants were RT-PCR positive for influenza at any time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
percentage of participants | 0.5 [0.01 to 2.65] | 2.6 [0.55 to 7.50]

12. Secondary Outcome: Mortality Rate at Day 28
Time Frame: Up to Day 28
Population: Participants were RT-PCR positive for influenza at any time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
percentage of participants | 1.9 [0.53 to 4.85] | 5.3 [1.96 to 11.10]

13. Secondary Outcome: Time to NEWS2 of ≤ 2 Maintained for 24 Hours
Description: A score of 0 (Range 0 - 3) indicates normal health conditions.
Time Frame: Up to Day 35
Population: Participants were RT-PCR positive for influenza at any time point
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 208 | 114
hours | 106.3 [88.3 to 138.3] | 127.2 [77.4 to 156.3]

14. Secondary Outcome: Time to Cessation of Viral Shedding by Virus Titer
Description: Time to cessation of viral shedding by virus titer is defined as the time, in hours, between the initiation of study treatment and first time when the influenza virus titer is below the limit of detection (0.75 log10 TCID50/mL)
Time Frame: Screening (baseline) and on Days 2, 3, 4, 5, 7, and 10
Population: Participants were RT-PCR positive for influenza at any time point and with a positive virus titer on Day 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 159 | 78
hours | 23.9 [23.2 to 24.5] | 63.7 [46.4 to 68.1]

15. Secondary Outcome: Change From Baseline in Influenza Virus Titer at Each Timepoint
Description: Influenza virus titer is the quantity of influenza virus in a given volume within the samples obtained from nasal swabs. If influenza virus titer was less than the lower limit of quantification, the virus titer was imputed as 0.749 (log10TCID50/mL). A lower value indicates lower viral titer.
Time Frame: Days 2, 3, 4, 5, 7, and 10
Population: Participants were RT-PCR positive for influenza at any time point and with a positive virus titer on Day 1
Measure: Number; unit: log10 TCID50/ml
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 159 | 78
log10 TCID50/ml
  Day 2: number analyzed (Participants) | 159 | 76
  Day 2 | -2.36 | -1.00
  Day 3: number analyzed (Participants) | 156 | 73
  Day 3 | -2.70 | -1.93
  Day 4: number analyzed (Participants) | 152 | 75
  Day 4 | -2.88 | -2.50
  Day 5: number analyzed (Participants) | 153 | 72
  Day 5 | -3.01 | -2.81
  Day 7: number analyzed (Participants) | 147 | 69
  Day 7 | -3.00 | -2.95
  Day 10: number analyzed (Participants) | 144 | 69
  Day 10 | -3.02 | -3.06

16. Secondary Outcome: Percentage of Participants With Positive Influenza Virus Titer at Each Timepoint
Description: Influenza virus titer is the quantity of influenza virus in a given volume within the samples obtained from nasal swabs. If influenza virus titer was less than the lower limit of quantification, the virus titer was imputed as 0.749 (log10 TCID50/mL). A lower value indicates lower viral titer.
Time Frame: Days 2, 3, 4, 5, 7, and 10
Population: Participants were RT-PCR positive for influenza at any time point and with a positive virus titer on Day 1.
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 159 | 78
percentage of participants
  Day 2: number analyzed (Participants) | 60 | 76
  Day 2 | 37.7 | 80.3
  Day 3: number analyzed (Participants) | 156 | 73
  Day 3 | 18.6 | 53.4
  Day 4: number analyzed (Participants) | 152 | 75
  Day 4 | 7.9 | 26.7
  Day 5: number analyzed (Participants) | 153 | 72
  Day 5 | 1.3 | 20.8
  Day 7: number analyzed (Participants) | 147 | 69
  Day 7 | 2.7 | 5.8
  Day 10: number analyzed (Participants) | 144 | 69
  Day 10 | 1.4 | 1.4

17. Secondary Outcome: Area Under the Curve in Virus Titer
Time Frame: Days 1, 2, 3, 4, 5, 7, and 10
Population: Participants with a positive virus titer on Day 1
Measure: Mean (Standard Deviation); unit: log10 TCID50/mL*hours
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 159 | 77
log10 TCID50/mL*hours | 291.68 (176.68) | 332.04 (183.63)

18. Secondary Outcome: Time to Cessation of Viral Shedding by RT-PCR
Description: Time to cessation of viral shedding by RT-PCR, in hours, is defined as the time between the initiation of study treatment and first time when the virus RNA by RT-PCR is below the limit of detection (2.05 for flu A and 2.83 for flu B log10 virus particles/mL)
Time Frame: Screening (baseline) and on Days 2, 3, 4, 5, 7, and 10
Population: Participants were RT-PCR positive for influenza on Day 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 205 | 111
hours | 216.3 [211.3 to 239.8] | 261.1 [236.4 to NA] — Due to low number of events the upper limit of the 95% confidence interval (CI) was not evaluable

19. Secondary Outcome: Change From Baseline in the Amount of Virus RNA (RT-PCR) at Each Timepoint
Description: If the amount of virus RNA was less than the lower limit of quantification, the amount of virus RNA was imputed as 2.18 for flu A and 2.93 for flu B (log10 virus particles/mL)
Time Frame: Days 2, 3, 4, 5, 7, and 10
Population: Participants were RT-PCR positive for influenza on Day 1
Measure: Number; unit: log10 virus particles/mL
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 205 | 111
log10 virus particles/mL
  Day 2: number analyzed (Participants) | 195 | 105
  Day 2 | -0.98 | -0.66
  Day 3: number analyzed (Participants) | 181 | 98
  Day 3 | -1.54 | -1.19
  Day 4: number analyzed (Participants) | 171 | 93
  Day 4 | -2.35 | -1.84
  Day 5: number analyzed (Participants) | 155 | 88
  Day 5 | -2.91 | -2.39
  Day 7: number analyzed (Participants) | 128 | 66
  Day 7 | -3.15 | -2.96
  Day 10: number analyzed (Participants) | 85 | 49
  Day 10 | -3.69 | -3.21

20. Secondary Outcome: Percentage of Participants Positive by RT-PCR at Each Timepoint
Description: as for outcome 19
Time Frame: Days 2, 3, 4, 5, 7, and 10
Population: Participants were RT-PCR positive for influenza on Day 1
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 205 | 111
percentage of participants
  Day 2: number analyzed (Participants) | 204 | 109
  Day 2 | 95.6 | 96.3
  Day 3: number analyzed (Participants) | 201 | 105
  Day 3 | 90.0 | 93.3
  Day 4: number analyzed (Participants) | 194 | 107
  Day 4 | 88.1 | 87.9
  Day 5: number analyzed (Participants) | 194 | 103
  Day 5 | 79.9 | 85.4
  Day 7: number analyzed (Participants) | 184 | 97
  Day 7 | 69.6 | 68.0
  Day 10: number analyzed (Participants) | 182 | 97
  Day 10 | 46.7 | 50.5

21. Secondary Outcome: Area Under the Curve in the Amount of Virus RNA (RT-PCR)
Time Frame: Days 1, 2, 3, 4, 5, 7, and 10
Population: Participants were RT-PCR positive for influenza on Day 1.
Measure: Mean (Standard Deviation); unit: log10 virus particles/mL*hours
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 197 | 106
log10 virus particles/mL*hours | 676.40 (371.72) | 740.15 (484.07)

22. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. A serious adverse event (SAE) is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/ incapacity, is a congenital anomaly/ birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: Up to Day 35
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 239 | 124
percentage of participants
  AEs | 45.2 | 50.0
  SAEs | 12.1 | 15.3

23. Secondary Outcome: Percentage of Participants With AEs and SAEs Leading to Discontinuation From Treatment
Description: Discontinuation from study treatment.
Time Frame: Up to Day 35
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 239 | 124
percentage of participants
  AEs | 1.3 | 3.2
  SAEs | 0.8 | 1.6

24. Secondary Outcome: Percentage of Participants With Any Post-Treatment ALT and AST Above Baseline and >3 × ULN, >5 × ULN, >10 × ULN
Description: ALT = alanine aminotransferase AST = aspartate transaminase
Time Frame: Up to Day 35
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo
Number analyzed (Participants) | 239 | 124
percentage of participants
  AST(U/L) or ALT (U/L) >3 x ULN | 4.6 | 8.9
  AST(U/L) or ALT (U/L) >5 x ULN | 0.8 | 3.2
  AST(U/L) or ALT (U/L) >10 x ULN | 0 | 1.6

25. Secondary Outcome: Plasma Concentration of Baloxavir (Active Metabolite) at Specified Time Points
Time Frame: Day 1, 2, 4, 5, 7 and 8
Population: Participants who provided informed consent to intensive PK sampling in the Baloxavir Marboxil arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 8
ng/mL
  Day 1 - 30 minutes postdose: number analyzed (Participants) | 7
  Day 1 - 30 minutes postdose | 37.82 (23.61)
  Day 1 - 2 hours postdose | 75.06 (52.16)
  Day 1 - 4 hours postdose | 95.85 (58.36)
  Day 1 - 10 hours postdose: number analyzed (Participants) | 7
  Day 1 - 10 hours postdose | 64.47 (39.47)
  Day 2 - 24 hours postdose | 53.36 (37.42)
  Day 4 - Predose | 24.26 (15.87)
  Day 4 - 30 minutes postdose | 49.16 (52.07)
  Day 4 - 2 hours postdose: number analyzed (Participants) | 5
  Day 4 - 2 hours postdose | 109.66 (95.22)
  Day 4 - 4 hours postdose | 117.69 (60.54)
  Day 4 - 10 hours postdose: number analyzed (Participants) | 5
  Day 4 - 10 hours postdose | 94.08 (49.71)
  Day 5 - 24 hours postdose | 77.98 (42.89)
  Day 7 - predose: number analyzed (Participants) | 5
  Day 7 - predose | 23.31 (25.87)
  Day 8 - 24 hours postdose: number analyzed (Participants) | 1
  Day 8 - 24 hours postdose | 105.00 (NA) — Not applicable as only 1 participant was analyzed
  Visit 8: number analyzed (Participants) | 6
  Visit 8 | 28.37 (61.61)

26. Secondary Outcome: Area Under the Concentration to Time Curve From Time 0 to 72 Hours (AUC0-72) of Baloxavir
Time Frame: 0, 0.5, 2, 4, 10, 24, 72 hours from dose on Day 1 and on Day 4, and Day 7, Day 8
Population: Participants who provided informed consent to intensive pharmacokinetic (PK) sampling in the Baloxavir Marboxil arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours(h)*nanogram(ng)/milliliter (mL)
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 8
Hours(h)*nanogram(ng)/milliliter (mL)
  Day 1 | 2820 (70.5)
  Day 4: number analyzed (Participants) | 5
  Day 4 | 3170 (53.5)
  Day 7: number analyzed (Participants) | 0
  Day 8: number analyzed (Participants) | 0

27. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Baloxavir
Time Frame: 0, 0.5, 2, 4, 10, 24, 72 hours from dose on Day 1 and on Day 4, and Day 7, Day 8
Population: Participants who provided informed consent to intensive PK sampling in the Baloxavir Marboxil arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 8
ng/mL
  Day 1 | 86.3 (64.6)
  Day 4 | 123 (51.7)
  Day 7: number analyzed (Participants) | 0
  Day 8: number analyzed (Participants) | 0

28. Secondary Outcome: Apparent Half-Life (T1/2) of Baloxavir
Time Frame: 0, 0.5, 2, 4, 10, 24, 72 hours from dose on Day 1 and on Day 4, and Day 7, Day 8
Population: Participants who provided informed consent to intensive PK sampling and had a sufficient number of samples available for analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 8
Hours (h)
  Day 1: number analyzed (Participants) | 1
  Day 1 | 18.9 (NA) — Not estimable as only 1 participant was eligible for the assessment of this measure
  Day 4: number analyzed (Participants) | 2
  Day 4 | 23.4 (12.8)
  Day 7: number analyzed (Participants) | 0
  Day 8: number analyzed (Participants) | 0

29. Secondary Outcome: Concentration at 24 Hours (C24) of Baloxavir
Time Frame: 0, 0.5, 2, 4, 10, 24, 72 hours from dose on Day 1 and on Day 4, and Day 7, Day 8
Population: Participants who provided informed consent to intensive PK sampling in the Baloxavir Marboxil arm
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Baloxavir Marboxil
Number analyzed (Participants) | 8
ng/mL
  Day 1 | 43.9 (74.4)
  Day 4 | 67.1 (66.8)
  Day 7: number analyzed (Participants) | 1
  Day 7 | 105 (NA) — Not applicable as only 1 participant was analyzed
  Day 8: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Randomization up to Day 35
Arm/Group | Baloxavir Marboxil | Placebo
All-Cause Mortality (participants affected / at risk) | 4/239 | 7/124
Serious Adverse Events (participants affected / at risk) | 29/239 | 19/124
Other Adverse Events (participants affected / at risk) | 44/239 | 27/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baloxavir Marboxil (N=239) | Placebo (N=124)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Graft versus host disease (Immune system disorders) | 0 (0) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 5 (5)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Superinfection viral (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baloxavir Marboxil (N=239) | Placebo (N=124)
Constipation (Gastrointestinal disorders) | 10 (10) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 6 (7)
Nausea (Gastrointestinal disorders) | 7 (9) | 4 (4)
Pneumonia (Infections and infestations) | 5 (6) | 4 (4)
Hepatic enzyme increased (Investigations) | 6 (7) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (9) | 5 (5)
Headache (Nervous system disorders) | 9 (11) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT03684044/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03684044/SAP_001.pdf